CLINICAL TRIAL: NCT02214810
Title: A Randomized, Single-blinded, Prospective Study of Postsurgical Pain Control After Open Reduction and Internal Fixation of Lower Extremity Fractures With Liposomal Marcaine.
Brief Title: A Study of Postsurgical Pain Control for Lower Extremity Fractures
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Broward Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5187
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Lower Extremity Fractures.
Keywords: Bupivacaine; multimodal; exparel; open reduction; internal fixation; post-surgical pain control
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control- Marcain (Active Comparator): Group 1 will receive non-liposomal bupivacaine introduced into the soft tissue surrounding the fracture at the conclusion of the surgery.
  Interventions: Drug: Bupivacaine/Exparel
- Experimental- Exparel (Experimental): Group 2 will receive a mixture of non-liposomal bupivacaine and Exparel introduced into the soft tissue surrounding the fracture at the conclusion of the surgery.
  Interventions: Drug: Bupivacaine/Exparel

INTERVENTIONS:
Drug: Bupivacaine/Exparel — The opaque envelope, which was selected by the treating physician, will accompany each of the study participants will be opened and the patient identified as belonging to either Group 1 or Group 2. It is important to note that randomization of the envelopes were computer-generated and placed by a co-investigator; the treating physician is completely unaware of the order of the opaque envelopes. Patients in Group 1 will receive a standardized medication regimen including non-liposomal bupivacaine by soft-tissue injection at the conclusion of their surgical procedure. Those in Group 2 will receive non-liposomal bupivacaine and ExparelTM by soft-tissue injection at the conclusion of their surgical procedure. Study participants will undergo injection in this manner until the conclusion of the study.

SUMMARY:
Postsurgical pain may effectively be treated with a multimodal approach that incorporates the use of local anesthetics. Bupivacaine is a local anesthetic that has been proven to be effective at reducing postsurgical pain. Furthermore, this local anesthetic has been shown to reduce opioid use, improve functional outcomes, allow for early mobilization, and decrease hospital length of stay. However, local anesthetics, via wound infiltration, are often short-acting and do not meet the duration of postsurgical pain due to their solubility and protein-binding properties. ExparelTM is an FDA-approved liposomal formulation of bupivacaine that allows for 72 hours of postsurgical analgesia with a single injection. This formulation has been shown to have little to no adverse effects; although some studies have reported adverse effects with the use of ExaprelTM, most frequently being nausea, vomiting, and dizziness. The occurrences of these adverse events were still less than the placebo cohort.

DETAILED DESCRIPTION:
All patients undergoing surgical fixation of a lower extremity fracture(s) will be offered the opportunity to enroll in the study. Patients undergoing unilateral or bilateral surgical fixation would be included. Written, informed consent to enrollment will be recorded and included in the patient record. The study is designed around the standard of care for postsurgical pain management. There are no additional costs to the patient strictly related to this study.

Patients will undergo surgical fixation of a lower extremity fracture(s) by one of surgical investigators at a single institution. A sealed, opaque envelope, selected in the pre-operative holding area, will accompany each patient participant to the operating room. The envelope will be opened at the conclusion of the fracture fixation to reveal patient assignment to either study Group 1 or Group 2. Once the total numbers of patients have completed their procedures and follow-up, the study will close.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Preoperative diagnosis of lower extremity fracture(s) requiring surgical fixation

Exclusion Criteria:

* Allergy to ExparelTM or certain other local anesthetic agents
* Surgery performed at an outside institution or by a different surgeon
* Chronic analgesic users (defined as use of opioid medication >14 days in the past 3 months, or use of non-opioid pain medication >5 times per week
* Pregnant females or females who think they may become pregnant
* Peripheral neuropathy
* Major psychiatric disease
* Inability to comprehend the nature of the study
* Unwillingness to provide signed informed consent
* Markedly abnormal kidney function or renal disease
* Non-English speaking
* Signs or symptoms of compartment syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Visual Analogue Scale (VAS) | 72 hours
  Patients will be asked to complete a Pain Visual Analogue Scale every 2 hours for the first 12 hours of their stay (2, 4, 6, 8, 10, 12), and then again at 24, 30 and 72 hours into their hospitalization.

SECONDARY OUTCOMES:
Pain Management Satisfaction | 2 weeks, post-operatively
  Patients will complete the post-surgery satisfaction form at their 2-week, post-operative office visit.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Cross, MD, Principal Investigator — Broward Health
Locations (1):
- Broward Health Medical Center, Fort Lauderdale, Florida, United States

REFERENCES:
- [Result] References 1-Candoitti 2012 2-Gupta Curr Opin Anaesthesiol 2010, Liu J Am Coll Surg 2006 3-Lynch Anesth Analg 1997, Amin J Surg Pakistan 2010 4-Golf Adv Ther 2011, Onel 2011, Bergese IARS Annual Meeting 2011 5-Angst Clin Pharmacokinet 2006, Howell Cancer J 2001